CLINICAL TRIAL: NCT00361062
Title: Aggressive Behavior Induced by SSRIs During the First Month of Treatment
Brief Title: Aggressive Behavior Induced by Selective Serotonin Reuptake Inhibitors (SSRIs) During the First Month of Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Dalya Navot-MIntzer, HaEmek Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: hae064910706ctil
Record Dates: First submitted 2006-08-04; First posted 2006-08-07 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Adverse Effects; Aggression
Keywords: aggressive; SSRI's; simulation; behavioral; Side Effects, Psychological; adverse effects; Serotonin Reuptake Inhibitors; aggressive behavior; computer simulation
MeSH Terms: conditions — Aggression; Behavior

INTERVENTIONS:
Behavioral: comparative computer simulation — comparative computer simulation assessing the level of aggressiveness before and after the beginning of SSRI treatment.

SUMMARY:
SSRIs are the first line of therapy for anxiety and depressive disorders and for many other clinical diagnoses. One of the most disturbing side effects that is observed is a tendency towards aggressiveness among patients receiving medications from this group, mainly during the first month of therapy. Aggressive behavior tends to occur in some individuals but not in others. In some sub-groups of people, personality and character traits might make a person more prone to aggressive behavior.

In this study the investigators try to estimate the tendency towards aggressive behavior in patients prescribed to a medication from the SSRI group. By using a comparative computer simulation they hope to be able to detect delicate changes and to maybe get some clues of the personalities prone to aggressive behavior in the future.

DETAILED DESCRIPTION:
Selective serotonin reuptake inhibitors (SSRIs) became the first line therapy for anxiety and depressive disorders and for many other clinical diagnoses. One of the most disturbing side effects that is observed is a tendency towards aggressiveness among patients receiving medications from this group, mainly during the first (one month) period of therapy. Aggressive behavior tends to occur in some individuals but not in others. Until now most of the cases and reports in the literature demonstrate the extreme events of aggressive behavior. These personality or any other character traits that are more prone to develop aggressiveness have not been studied and it is not clear if this side effect manifests itself just in the extreme rare cases or if it is a more common phenomenon that occurs in a wider group of people.

In this study we try to estimate the tendency towards aggressive behavior of patients prescribed to a medication of the SSRI group. By using a comparative computer simulation we hope to be able to detect more delicate changes and maybe to get some clues of the personalities prone to aggressive behavior in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Instructed by his/her family physician to start taking a medicine in the SSRI group

Exclusion Criteria:

* According to the family practitioner's record: under SSRI, SNRI, or NRI treatment during the previous 3 months or at the time of entry into the study.
* Diagnosed with schizophrenia or active psychosis or impaired judgment
* Anti-social personality disorder
* Drug use or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-09 (Actual); Primary Completion 2008-07 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
aggressiveness level | whithin 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Dalya Navot-Mintzer, MD, Principal Investigator — HaEmek Medical Center, Family Practice Ward; Dalya Navot-Mintzer, MD, Study Director — HaEmek Medical Center, Family Practice Ward
Locations (2):
- Israel (2):
  - HaEmek Medical Center, Afula, Ysrael Valley
  - HaEmek Medical Center, Afula